CLINICAL TRIAL: NCT02374580
Title: Partnership and Dignity: a Mixed-methods Survey on Supporting and Retaining Uganda's Village Health Teams
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: VHT_041406
Record Dates: First submitted 2014-12-04; First posted 2015-03-02 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2015-08

CONDITIONS: Malaria; Diarrhea; Pneumonia
MeSH Terms: conditions — Malaria; Diarrhea; Pneumonia

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
For more than a decade, Uganda's Ministry of Health has led a community health worker program model in which Village Health Teams (VHTs), cadres of unpaid volunteers, are assigned the task of delivering preventative health services and education to their local communities. Studies have demonstrated the effectiveness of Uganda's VHTs in improving certain health outcomes; however it is known that VHTs are not optimally supported, and there has been VHT attrition in recent years. The Ministry of Health has recognized the inadequate support of VHTs thus far and is aiming to "expand VHTs to all local governments and explore ways of sustaining VHTs." The objective of this study is to evaluate the extent to which material support is a deciding factor in the efficiency and durability of Uganda's VHT initiative. Material support may take the form of monetary stipends, regular payment, transportation assistance, or nonfinancial materials such as bicycles or mobile phone airtime. This study will review existing literature and gather novel data through surveys of VHT members and VHT stakeholders. The quantitative and qualitative survey data will be analyzed for trends that may point to a conclusion in the context of existing health policy discourse on community health worker remuneration. The purpose of this study is to strengthen the knowledge base on whether or not the current absence of material support significantly limits the potential for Uganda's VHTs to be sustained and expanded. This information can be used by governmental and non-governmental organizations in their work to strengthen and sustain VHTs throughout the country.

ELIGIBILITY:
Inclusion Criteria:

VHT subjects must have been actively working as a VHT member for at least 6 months. Stakeholders, that is, program managers, health administrators and policy makers, must be involved in managing, administrating, or guiding policy for VHT programs as part of their official job description. These persons must also have been acting in those roles for at least 6 months. All study subjects will be 18 years of age or older. All study subjects will be literate and able to be informed to give or withhold consent of participation.

Exclusion Criteria:

There will be no exclusion or inclusion based on gender, race, tribal or ethnic affiliation, religion, or health status.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of at least 200 individual working VHT members, and at least 10 stakeholders, that is, program managers, administrators, district health officers, and policymakers. Almost all study subjects will be of Ugandan nationality. Some stakeholders may be expatriates.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2015-02; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Predicted longevity related to support sufficiency | Up to 5 months
  This outcome will be measured by asking VHTs to rate aspects of their current support. We will follow up those questions by asking how long they expect to be able to continue in their position as VHTs. The two results will be evaluated for possible trends connecting sufficiency of existing support with predicted longevity.

SECONDARY OUTCOMES:
Predicted longevity of minimum 10 years if current support does not increase | Up to 5 months
  This outcome will be measured by asking the VHTs if they predict being able to continue in their positions for at least 10 more years if their current support does not increase.

CONTACTS AND LOCATIONS:
Overall Officials: William S Schroth, MD MPH, Principal Investigator — George Washington University School of Medicine and Health Sciences
Locations (1):
- The George Washington University School of Medicine and Health Sciences, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Ministry of Health, Uganda, Education and Promotion Division. Village health team strategy and operational guidelines. 2010.
- [Background] Brenner JL, Kabakyenga J, Kyomuhangi T, Wotton KA, Pim C, Ntaro M, Bagenda FN, Gad NR, Godel J, Kayizzi J, McMillan D, Mulogo E, Nettel-Aguirre A, Singhal N. Can volunteer community health workers decrease child morbidity and mortality in southwestern Uganda? An impact evaluation. PLoS One. 2011;6(12):e27997. doi: 10.1371/journal.pone.0027997. Epub 2011 Dec 14. PMID 22194801
- [Background] Okello D, Floyd K, Adatu F, Odeke R, Gargioni G. Cost and cost-effectiveness of community-based care for tuberculosis patients in rural Uganda. Int J Tuberc Lung Dis. 2003 Sep;7(9 Suppl 1):S72-9. PMID 12971657
- [Background] Kalyango JN, Rutebemberwa E, Alfven T, Ssali S, Peterson S, Karamagi C. Performance of community health workers under integrated community case management of childhood illnesses in eastern Uganda. Malar J. 2012 Aug 20;11:282. doi: 10.1186/1475-2875-11-282. PMID 22905758
- [Background] Kayemba Nalwadda C, Guwatudde D, Waiswa P, Kiguli J, Namazzi G, Namutumba S, Tomson G, Peterson S. Community health workers - a resource for identification and referral of sick newborns in rural Uganda. Trop Med Int Health. 2013 Jul;18(7):898-906. doi: 10.1111/tmi.12106. Epub 2013 Apr 2. PMID 23551394
- [Background] Ministry of Health Uganda. Annual Health Sector Performance Report: Financial Year 2012/2013. 2013.
- [Background] Ministry of Health Uganda. The second national health policy. 2010.
- [Background] Perry, H, et al. How effective are community health workers? an overview of current evidence with recommendations for strengthening community health worker programs to accelerate progress in achieving the health-related millennium development goals. Johns Hopkins University Bloomberg School of Public Health. 2012.
- [Background] Lehmann U., Sanders D. Community health workers: what do we know about them? The state of the evidence on programmes, activities, costs and impact on health outcomes of using community health workers. (2007) Geneva: World Health Organization. Available at: <http://www.who.int/hrh/documents/community_health_ workers.pdf>